CLINICAL TRIAL: NCT04773262
Title: Submaximal Cardiopulmonary Exercise Testing in Patients With Knee Osteoarthritis Scheduled for Total Knee Arthroplasty: a Feasibility Study
Brief Title: Feasibility of CPET in Patients Prior to TKA
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Anna hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NL76561.068.21
Record Dates: First submitted 2021-01-29; First posted 2021-02-26 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2021-02

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee; Cardiopulmonary Exercise Testing; Feasibility
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Higher aerobic capacity before surgery, as indicated during submaximal exercise testing by the oxygen uptake (VO2) at the ventilatory anaerobic threshold (VAT), is assumed to be prognostic for a better and faster postoperative recovery in patients with knee osteoarthritis (OA) undergoing total knee arthroplasty (TKA). Cardiopulmonary exercise testing (CPET) is the gold standard to measure aerobic capacity; however, it is unclear whether it is feasible to perform CPET using cycle ergometry in patients with knee OA prior to TKA surgery. The hypothesis is that performing CPET is feasible and participants will meet the feasibility criteria for success.

The primary objective of this cross-sectional feasibility study is to investigate the feasibility of CPET in patients with knee OA three to six weeks prior to TKA surgery in three domains: a) recruitment rate of participants who are representative of the target study population; b) reaching the VAT during CPET; and c) acceptability and suitability. The secondary objective is to investigate aerobic capacity of the study population and to compare values with normative values.

The study population consists of patients with knee OA scheduled for primary unilateral TKA surgery.

Feasibility of CPET will be assessed against five criteria: 1) recruitment rate ≥20%; 2) CPET performance rate ≥90%; 3) ≥90% of participants reached the VAT; 4) no serious adverse events; and 5) ≥80% of participants had a positive attitude towards CPET. Aerobic capacity is determined by the VO2 at the VAT and the oxygen uptake efficiency slope (OUES).

CPET is considered a safe procedure. Participants perform the CPET instead of a walking test following the standard preoperative screening and complete a questionnaire to examine their experiences. The investigator will contact the participants one week after the CPET to inquire whether they have developed any complaints afterwards. Benefit from participation is that all patients objectively get insight in their preoperative aerobic capacity.

DETAILED DESCRIPTION:
It is unclear whether it is feasible to perform submaximal exercise testing using cycle ergometry to measure aerobic capacity in patients with knee osteoarthritis (OA) undergoing total knee arthroplasty (TKA). Individuals prior to TKA surgery experience increasing knee pain and are progressively restricted in their activities of daily living (ADL), sports and work, which negatively affect their aerobic capacity. This causes severe deconditioning, which is more prominent in patients with more severe knee OA. As part of usual care before TKA procedure, patients are screened for risk factors for delayed recovery by measuring physical functioning. Although various practical performance-based tests are performed, measuring aerobic capacity is included nowhere. Therefore, a walking test will be replaced by cardiopulmonary exercise testing (CPET) using cycle ergometry, which is the gold standard for measuring aerobic capacity.

A higher aerobic capacity prior to TKA surgery is assumed to be prognostic for a better and faster postoperative recovery. The first step is to explore whether it is feasible to perform a submaximal CPET prior to TKA surgery using cycle ergometry in patients with knee OA. When the feasibility criteria are met, the possible prognostic value of preoperative aerobic capacity on postoperative recovery can be investigated in a subsequent prospective cohort study.

Primary objective: to investigate the feasibility of submaximal CPET in patients with knee OA three to six weeks prior to TKA surgery in the MUMC+ and Anna Hospital regarding three domains: 1) recruitment rate of participants who are representative of the target study population; 2) feasibility of CPET procedure; and 3) acceptability and suitability of CPET. These domains are operationalized with five feasibility criteria.

Secondary objective: to explore the aerobic capacity of the study population, individuals with knee OA scheduled for TKA surgery, using submaximal parameters (VO2 at the VAT and OUES) and compare their aerobic capacity with normative values.

This cross-sectional study will be conducted at the Maastricht University Medical Center (MUMC+) and Anna Hospital. CPET will be performed three to six weeks before the TKA surgery following the preoperative screening. The study will include 15 to 20 participants.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for primary unilateral TKA surgery in MUMC+ or Anna Hospital;
* Diagnosis of OA;
* CPET can be performed three to six weeks before TKA surgery following the preoperative screening;
* Mastery of the Dutch language.

Exclusion Criteria:

* Undergoing revision arthroplasty, bilateral TKA or hemi-arthroplasty surgery;
* Contraindications for CPET according to the American Thoracic Society (ATS) Statement on CPET and following the American Heart Association/American College of Sports Medicine (AHA/ACSM) Health/Fitness facility pre-participation screening questionnaire;
* Unable to get on and off a stationary bike;
* Complete dependence on a wheelchair;
* Serious comorbidities (e.g. malignancy, stroke);
* Cognitive impairments;
* Unable to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be included from the preoperative assessment clinic for TKA at the department of Physical Therapy at the MUMC+ and Anna Hospital with a diagnosis of symptomatic end-stage OA of the knee. It was decided to undergo an unilateral primary TKA surgery, because of failing of conservative treatment(s) and/or worsening of knee complaints.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of CPET | Item 1 through study completion, an average of 9 months; items 2-4 immediately after CPET performance; and item 5 within one week after CPET performance.
  Feasibility criteria:
  1. recruitment rate ≥20%: the percentage of eligible patients who gave informed consent to participate in the study;
  2. CPET performance rate ≥90%: the percentage of recruited participants actually performing CPET. They were able to pedal the bicycle around with 60 revolutions per minute (rpm) and cycling was not hindered by restricted knee flexion;
  3. ≥90% of participants reached the VAT (success rate): the percentage of participants who reached the VO2 at the VAT during CPET performance;
  4. 0% of participants experience serious adverse events during or after the test; and
  5. ≥80% of participants had a positive attitude towards CPET: the percentage of participants who are willing to perform the exercise test again at a later moment.

SECONDARY OUTCOMES:
Aerobic capacity: oxygen uptake (VO2) at the ventilatory anaerobic threshold (VAT), absolute value | Immediately after CPET performance.
  VO2 at the VAT in ml min-1.
Aerobic capacity: oxygen uptake (VO2) at the ventilatory anaerobic threshold (VAT), relative value | Immediately after CPET performance.
  VO2 at the VAT in ml kg-1 min-1.
Aerobic capacity: oxygen uptake efficiency slope (OUES), absolute value | Immediately after CPET performance.
  OUES; using all test data.
Aerobic capacity: oxygen uptake efficiency slope (OUES), normalised for body mass | Immediately after CPET performance.
  OUES.kg-1; using all test data.

CONTACTS AND LOCATIONS:
Overall Officials: A.F. Lenssen, prof. dr., Principal Investigator — Department of physical therapy, Maastricht University Medical Center+ (MUMC+)
Locations (1):
- Maastricht UMC, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
Once the feasibility study is published and the research team decide to proceed with a subsequent prospective cohort study to investigate the possible prognostic value of preoperative aerobic capacity on postoperative recovery, the data will not yet be accessible. However, data will be made available for inspection after completion of the study. For verification, data will be made available for people who have the necessary permissions/rights.

REFERENCES:
- [Background] Philbin EF, Ries MD, French TS. Feasibility of maximal cardiopulmonary exercise testing in patients with end-stage arthritis of the hip and knee prior to total joint arthroplasty. Chest. 1995 Jul;108(1):174-81. doi: 10.1378/chest.108.1.174. PMID 7606955
- [Background] Philbin EF, Groff GD, Ries MD, Miller TE. Cardiovascular fitness and health in patients with end-stage osteoarthritis. Arthritis Rheum. 1995 Jun;38(6):799-805. doi: 10.1002/art.1780380613. PMID 7779123
- [Background] Ries MD, Philbin EF, Groff GD. Relationship between severity of gonarthrosis and cardiovascular fitness. Clin Orthop Relat Res. 1995 Apr;(313):169-76. PMID 7641476
- [Background] Ries MD, Philbin EF, Groff GD, Sheesley KA, Richman JA, Lynch F Jr. Improvement in cardiovascular fitness after total knee arthroplasty. J Bone Joint Surg Am. 1996 Nov;78(11):1696-701. doi: 10.2106/00004623-199611000-00009. PMID 8934484
- [Background] Orsmond GI, Cohn ES. The Distinctive Features of a Feasibility Study: Objectives and Guiding Questions. OTJR (Thorofare N J). 2015 Jul;35(3):169-77. doi: 10.1177/1539449215578649. PMID 26594739